CLINICAL TRIAL: NCT05521880
Title: Anchoring Intermittent Long Acting Antimicrobials to Medication for Opioid Use Disorder Treatment to Facilitate Structured Transitions of Care for People Who Use Drugs Admitted to the Hospital With Invasive Infections
Brief Title: Anchoring Sequential Intermittent Long Acting Antimicrobials With Medication for Opioid Use Disorder (MOUD) for Invasive Infections Related to Opioid Use
Acronym: AIM-STOP
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was not able to enroll adequate participants within predetermined timelines
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Shivakumar Narayanan, Asst Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00101580
Record Dates: First submitted 2022-08-22; First posted 2022-08-30 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Substance Use Disorders; Infection, Soft Tissue; Bacteremia; Osteomyelitis Acute; Septic Arthritis
Keywords: OPAT; oritavancin
MeSH Terms: conditions — Substance-Related Disorders; Soft Tissue Infections; Bacteremia; Arthritis, Infectious | interventions — oritavancin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Historical outcomes with standard of care treatment (Other): Historical outcomes with standard of care treatment involving IV antibiotics administered in a skilled nursing facility will be compared
  Interventions: Drug: Oritavancin

INTERVENTIONS:
Drug: Oritavancin — Sequential therapy with weekly doses of oritavancin 1200 mg in stable, discharge appropriate patients with opioid use related invasive infections collocated in setting of treatment for opioid use disorder

SUMMARY:
Standard of care for patients with opioid use disorder and complicated infections is discharge to subacute nursing facilities on IV antibiotics until completion of treatment course. We aim to determine the efficacy of an alternative strategy using intermittent outpatient oritavancin therapy dosed weekly combined with initiation and continuation of medication assisted treatment for opioid use disorder for completion of antimicrobial therapy in a 12 week prospective, open-label study. Patients hospitalized for a drug use related infection and thought to need prolonged parenteral antimicrobial therapy will be assessed by a substance use consultant and Infectious Diseases service. If they are not on Medication for Opioid Use Disorder (MOUD), they will be assessed for initiation of MOUD. A collaborative multidisciplinary discharge planning process will be initiated and will involve linkage to care. If they have an infection with a gram positive organism, and are thought to be clinically stable for hospital discharge, they will be assessed for appropriateness for oritavancin and first dose will be administered prior to discharge. They will have an intake into an opioid treatment program where they can access collocated services and will be discharged with linkage to care through a peer recovery coach. They will be assessed in this collocated clinic post discharge for optimization of MOUD and progress of infection and subsequent dose/s of oritavancin will be administered. Patients will be followed for 12 weeks for cure/completion of therapy and MOUD outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old
* Able and willing to sign consent
* Ongoing opioid use defined by self report of use of non prescription opioids within 3 months of hospitalization
* Has infection determined to be from opioid/drug use and needed prolonged parenteral antimicrobial therapy
* Gram positive organism as causal pathogen and expected to be sensitive to oritavancin
* Deemed to be clinically stable for discharge (i.e no need for surgical intervention, with stable vital signs,afebrile and bacteremia cleared if present at admission for at least 72 hours)
* Not on opioid agonist therapy at admission to hospital and willing to initiate medication for opioid use disorder, which includes methadone/suboxone
* Willing and able to follow up for MOUD in colocated clinic site
* If female, the patient is surgically sterile, postmenopausal, or, if of childbearing potential, agrees to use at least 2 highly effective methods of birth control (e.g. prescription oral contraceptives, contraceptive injections, contraceptive patch, intrauterine device, barrier methods, abstinence) for the duration of the study until 60 days after study drug administration, or male partner sterilization alone

Exclusion Criteria:

* Known immediate hypersensitivity to oritavancin or glycopeptides
* Decompensated liver disease (Childs Pugh B or C) or Stage IV/V chronic kidney disease or acute kidney injury with creatinine clearance <30
* Unable to comply with research study visits
* Poor venous access not allowing screening laboratory collection
* Have any condition that the investigator considers a contraindication to study participation
* Pregnant or breastfeeding woman
* Require valve replacement surgery or have prosthetic material in body including prosthetic joints or non bioprosthetic valves.
* Polymicrobial infection
* Multisite infection- defined as >2 different organ system involvement or non-contiguous sites of same organ system which may need different duration of antimicrobial therapy.
* Lack of source control i.e lack of drainage of infected fluid collections, debridement of infected solid or necrotic tissue, removal of devices or foreign bodies, or definitive measures to correct anatomic derangements resulting in ongoing microbial contamination. This will be determined by investigator.
* Need for subacute rehabilitation due to physical frailty either chronic, or from hospitalization.
* Acute stroke during hospitalization.
* Severe neutropenia- ANC <500 or thrombocytopenia - platelet count <50,000.
* On prohibited concomitant medications

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-05-22 (Actual); Study Completion 2025-05-23 (Actual)

PRIMARY OUTCOMES:
Frequency of clinically assessed cure, completion (no need for further parenteral antimicrobial therapy) or transition to suppressive antimicrobial therapy at 12 weeks for patients discharged to home with long acting agents and MOUD | 12 weeks

SECONDARY OUTCOMES:
Frequency of non-adherence to antimicrobial therapy (lack of follow up or any subsequent scheduled parenteral antimicrobial dose administration) | 12 weeks
Frequency of hospital readmission at 30 days post discharge and at 90 days post discharge | 12 weeks
Proportion of patients with drug related AE | 12 weeks
Rate of follow up at scheduled in person Medication for Opioid Use Disorder (MOUD) visit and frequency of follow up/no shows at follow up dosing visits for MOUD at 12 weeks | 12 weeks
Proportion of patients with positive urine drug screen | 12 weeks
Evaluate effect of Medication for Opioid Use Disorder (MOUD) follow up on cure/completion or transition to suppressive antimicrobial therapy. | 12 weeks
Rate of direct acting antiviral (DAA) initiation for Hepatitis C (HCV) in patients enrolled and rate of DAA completion and SVR for HCV in patients enrolled | 6 months

OTHER OUTCOMES:
Rates of new HIV infection | 12 weeks
Rates of occurrence of new bacterial infection related to OUD | 12 weeks
Rates of high risk behavior at baseline and during and post completion of antimicrobial therapy and follow up. | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided